CLINICAL TRIAL: NCT06700317
Title: Intraoperative Hyperspectral Imaging for Laparoscopic Surgery (LapHSI): a Multicentre Post-market Clinical Study
Brief Title: Intraoperative Hyperspectral Imaging for Laparoscopic Surgery
Acronym: LapHSI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 321001
Record Dates: First submitted 2024-11-20; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Neoplasms; Colorectal Surgery; Cholecystitis; Cholecystectomy, Laparoscopic
Keywords: hyperspectral imaging; surgery; laparoscopic surgery; colorectal cancer; cholecystitis
MeSH Terms: conditions — Colorectal Neoplasms; Cholecystitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HSS1 (Experimental): Surgery performed using HSS1
  Interventions: Device: HSS1

INTERVENTIONS:
Device: HSS1 — Surgery performed using HSS1

SUMMARY:
The study aims to evaluate the use of the HyperSnap Surgical System (HSS1) during laparoscopic surgeries, specifically in bowel resections and cholecystectomies.

DETAILED DESCRIPTION:
The study will observe patients undergoing bowel resection and cholecystectomy surgeries to determine if HyperSnap Surgical System (HSS1), as a primary visualisation tool, functions safely and capably as a laparoscopic imager. In addition, we will see if it subjectively improves the identification of critical anatomical structures. In addition, the study will secondarily assess how StO2 information may be included in the surgical workflow and how surgeons may react to this additional information.

ELIGIBILITY:
Inclusion Criteria:

A) Cholelithiasis or cholecystitis with indications for laparoscopic surgery (cholecystectomy)

* Adult patients aged 18 years and over
* Common bile duct diameter < 8mm as assessed using ultrasound
* Patients able to provide written informed consent

B) Colorectal cancer requiring elective bowel resection via a laparoscopic approach.

* Adult patients aged 18 years and over
* Patients who are scheduled for elective laparoscopic colon cancer resection
* Patients able to provide written informed consent

Exclusion Criteria:

A) Cholelithiasis or cholecystitis with indications for laparoscopic surgery (cholecystectomy)

* Patients under 18 years of age
* Patients with a history of previous abdominal surgery and multiply scarred abdomen
* Common bile duct diameter ≥ 8mm as assessed using ultrasound
* Patients unable to provide written informed consent
* Patients who are pregnant

B) Colorectal cancer requiring elective bowel resection via a laparoscopic approach.

* Patients under 18 years of age
* Patients with a history of previous abdominal surgery and multiply scarred abdomen
* Patients unable to provide written informed consent
* Patients undergoing emergency surgery
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Device safety | From enrollment to end of follow up (30 days)
  To demonstrate that under normal conditions of use, the performance characteristics of the device are those intended, enabling laparoscopic abdominal surgery to be safely performed using the UKCA-marked medical device (HSS1) as the primary surgical visualisation system.

SECONDARY OUTCOMES:
Technological performance | Duration of surgery
  To determine any undesirable side effects in technological performance and assess whether these constitute risks when weighed against the intended performance of the device.
Utility and usability of tissue oxygenation saturation maps in bowel surgery | Duration of surgery
  To assess the utility and usability of tissue oxygen saturation maps in bowel resection surgery for delineation of intestinal angiosomes and how the additional StO2 biomarker influenced clinical decision making
Utility and usability of tissue oxygenation saturation maps in cholecystectomy | Duration of surgery
  To perform retrospective analysis of the utility and usability of tissue oxygen saturation maps in cholecystectomy (not shown during procedure) for delineation of relevant anatomical structures within the surgical field.
Human factors analysis on use of HSS1 | Duration of surgery
  To perform a human factor analysis of the use of the UKCA marked medical device (HSS1) in relation to surgical workflow and surgeon performance.

IPD SHARING:
Plan to Share IPD: No